CLINICAL TRIAL: NCT06685601
Title: An Intervention Study on Transcranial Photobiomodulation for Children With Attention-Deficit/Hyperactivity Disorder
Brief Title: An Intervention Study on Transcranial Photobiomodulation in Children With Attention Deficit Hyperactivity Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Capital Medical University (Other); Peking Union Medical College (Other); Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QL000005
Record Dates: First submitted 2024-11-05; First posted 2024-11-12 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: ADHD - Attention Deficit Disorder With Hyperactivity
Keywords: tPBM; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active stimulation (Active Comparator): During the active stimulation condition, participants will receive a single session of tPBM intervention, lasting 12 minutes.
  Interventions: Device: tPBM（active）
- sham stimulation (Sham Comparator): During the sham stimulation condition, participants will receive the same intervention with identical target areas and wavelength, but only for the first and last 30 seconds of the session.
  Interventions: Device: tPBM（sham）

INTERVENTIONS:
Device: tPBM（active） — During the active stimulation condition, participants will receive a single session of tPBM intervention, lasting 12 minutes.
  Arms: active stimulation
Device: tPBM（sham） — During the sham stimulation condition, participants will receive the same intervention with identical target areas and wavelength, but only for the first and last 30 seconds of the session.
  Arms: sham stimulation

SUMMARY:
This study aims to intervene in children and adolescents with ADHD using transcranial photobiomodulation, comparing its effects on executive function at the levels of electroencephalography (EEG), eye tracking, and cognitive behavior. The goal is to identify the most effective clinical treatment strategy for ADHD patients.

DETAILED DESCRIPTION:
This study is conducted as a randomized triple-blind trial to investigate the effects of photobiomodulation therapy on ADHD. Initially, standardized assessment tools (physician ratings and parent self-reports) are employed to evaluate baseline clinical symptoms in ADHD patients who meet the inclusion and exclusion criteria. The experiment utilizes a within-subject design (within-subject factors: active versus sham stimulation), with each participant randomly assigned to receive two interventions-one active and one sham stimulation-administered in a counterbalanced order, with at least a one-week interval between the two sessions. Immediately following the intervention, standardized assessment tools are used to evaluate multidimensional clinical symptoms, and data related to executive function, including cognitive behavioral data, electroencephalographic data, and eye-tracking data, are collected. The intervention is carried out by trained technicians in accordance with the randomization results, while maintaining blinding for both clinical evaluators and participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 6 and 18 years;
2. Clinically diagnosed with ADHD by a psychiatrist;
3. Confirmed by the researcher (child psychiatrist) to meet the diagnostic criteria for Attention-Deficit/Hyperactivity Disorder as outlined in the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5);
4. M.I.N.I. KID interview shows only ADHD, with no other comorbidities;
5. Able to cooperate with transcranial photobiomodulation.
6. The participant and their guardian fully understand the study procedures and content and agree to participate in the study, signing the informed consent form.

Exclusion Criteria:

1. Diagnosis of other severe mental illnesses, such as schizophrenia or bipolar disorder;
2. Presence of severe physical diseases or conditions, such as significant intracranial lesions, thyroid disorders, epilepsy, congenital heart disease, severe hematologic disorders, systemic lupus erythematosus, auditory or visual impairments, etc.;
3. Presence of significant structural brain abnormalities on imaging studies;
4. Presence of severe neurological diseases with a clear family history or potential risk;
5. Presence of metal implants or a pacemaker, or holes or fractures in the skull;
6. Currently undergoing other ADHD treatments (e.g., methylphenidate or other pharmacological treatments, behavioral therapy, etc.) or has discontinued such treatments for less than 2 weeks;
7. Raven's Progressive Matrices IQ score < 85.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
EEG(Electroencephalogram) | From enrollment to the end of treatment at 3 weeks"
  The Electroencephalogram was recorded while participants performed a continuous attention task. The Negative 2-Posterior Contralateral(N2pc) waveform was analyzed, and a comparison of the N2pc waveforms following true and false stimuli was made to assess the improvement of attention in participants induced by transcranial light biofeedback.
Executive Function Task | From enrollment to the end of treatment at 3 weeks"
  Participants completed an executive function task following active and sham stimuli to compare the effects of transcranial Photobiomodulation on the improvement of executive function in children with ADHD.

SECONDARY OUTCOMES:
Swanson, Nolan, and Pelham Version IV | From enrollment to the end of treatment at 3 weeks"
  Participants completed the Swanson, Nolan, and Pelham Version IV (SNAP-IV) scale following active and sham stimuli to compare the effects of transcranial light biofeedback on the improvement of attention and hyperactivity-impulsivity symptoms in children with ADHD.
Sleep Disturbances Scale for Children | From enrollment to the end of treatment at 3 weeks"
  Participants completed the Sleep Disturbances Scale for Children (SDSC) scale following active and sham stimuli to compare the effects of transcranial Photobiomodulation on the improvement of sleep symptoms in children with ADHD.
Behavior Rating Inventory of Executive Function | From enrollment to the end of treatment at 3 weeks"
  Participants completed the Behavior Rating Inventory of Executive Function (BRIEF) scale following active and sham stimuli to compare the effects of transcranial Photobiomodulation on the improvement of attention control, emotional regulation, and behavioral inhibition in children with ADHD.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided